CLINICAL TRIAL: NCT02324465
Title: King Vision Video Laryngoscope Versus Glidescope Video Laryngoscope: A Comparative Study in Ambulatory Surgery Center Patients
Brief Title: King Vision Video Laryngoscope Versus Glidescope Video Laryngoscope
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to low enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Doug Hester, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 130470
Record Dates: First submitted 2014-12-18; First posted 2014-12-24 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- King Vision Video Laryngoscope (Active Comparator): The patient would be randomized to intubation via use of the King Vision VL
  Interventions: Device: King Vision Video Laryngoscope
- Glidescope Video Laryngoscope (Active Comparator): The patient would be randomized to intubation via use of the Glidescope VL
  Interventions: Device: Glidescope Video Laryngoscope

INTERVENTIONS:
Device: King Vision Video Laryngoscope — Intubation via King Vision Video Laryngoscope
  Other Names: King Systems
  Arms: King Vision Video Laryngoscope
Device: Glidescope Video Laryngoscope — Intubation via Glidescope Video Laryngoscope
  Other Names: Verathon
  Arms: Glidescope Video Laryngoscope

SUMMARY:
The investigators plan to conduct a randomized trial comparing the intubation success rate and time of the King Vision Video Laryngoscope to the Glidescope video laryngoscope in order to demonstrate the comparability of the devices.

DETAILED DESCRIPTION:
Both the King Vision and Glidescope video laryngoscopes are advanced airway devices that are relatively low cost and are designed to improve the efficiency of both routine and difficult intubation. Both systems use disposable blades, which eliminates the need for blade sterilization and may minimize the risk of infectious exposure to patients and improve cost and efficiency associated with the sterilization processing of non-disposable laryngoscopes. The Glidescope has been commercially available longer than the King Vision, and has been more frequently studied.

Although similar in many respects, the King Vision and Glidescope systems have differing designs which may result in differences in speed and success in the management of routine and/or difficult airways.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective, ambulatory surgery requiring general anesthesia and endotracheal intubation

Exclusion Criteria:

* Patients who require rapid sequence induction and intubation or fiberoptic intubation.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hester, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- King Vision Video Laryngoscope: The patient would be randomized to intubation via use of the King Vision VL then Glidescope VL
  King Vision Video Laryngoscope: Intubation via King Vision Video Laryngoscope
  Glidescope Video Laryngoscope: Intubation via Glidescope Video Laryngoscope
- Glidescope Video Laryngoscope: The patient would be randomized to intubation via use of the Glidescope VL then King Vision VL
  King Vision Video Laryngoscope: Intubation via King Vision Video Laryngoscope
  Glidescope Video Laryngoscope: Intubation via Glidescope Video Laryngoscope
Period: Overall Study
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope
Started | 18 | 22
Completed | 18 | 21
Not Completed | 0 | 1
Not completed — device failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 33
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Time Until Intubation With Each Device
Description: time from the introduction of the laryngoscope into the oral cavity to endotracheal tube reaching the glottic aperture
Time Frame: <100 seconds
Measure: Mean (Full Range); unit: seconds
Groups:
- King Vision Video Laryngoscope: The patient would be randomized to intubation via use of the King Vision VL or Glidescope VL
  King Vision Video Laryngoscope: Intubation via King Vision Video Laryngoscope
- Glidescope Video Laryngoscope: The patient would be randomized to intubation via use of the Glidescope VL or King Vision VL
  Glidescope Video Laryngoscope: Intubation via Glidescope Video Laryngoscope
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope
Number analyzed (Participants) | 18 | 21
seconds | 32.3 [10.0 to 69.7] | 27.2 [9.6 to 53.2]

2. Secondary Outcome: Mean Pulse Oximetry Saturation Value Reading During Intubation
Time Frame: <100 seconds
Measure: Mean (Full Range); unit: percentage of oxygen saturation
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope
Number analyzed (Participants) | 18 | 21
percentage of oxygen saturation | 97.39 [85 to 100] | 97.0 [82 to 100]

3. Secondary Outcome: Total Number of Assisted Maneuvers Required to Complete Intubation (Includes All Participants in Arm)
Description: Assisted Maneuvers can include laryngeal manipulation, head lift, Backward Upward Rightward Pressure, stylet removed, Cricoid pressure, scope manipulation and bougie.
Time Frame: <100 seconds
Measure: Number; unit: assisted maneuvers
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope
Number analyzed (Participants) | 18 | 21
assisted maneuvers
  Backward Upward Rightward Pressure | 0 | 1
  stylet removed | 0 | 1
  Cricoid pressure | 0 | 3
  bougie | 0 | 1
  scope manipulation | 0 | 1

4. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Notation of any injury to lips, teeth, soft tissue.
Time Frame: during and immediately after procedure (approx 180 minutes)
Measure: Number; unit: participants
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope
Number analyzed (Participants) | 18 | 22
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: approximately 180 minutes
Arm/Group | King Vision Video Laryngoscope | Glidescope Video Laryngoscope
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 2/18 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | King Vision Video Laryngoscope (N=18) | Glidescope Video Laryngoscope (N=22)
Lip Trauma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) — minor lacerations associated with intubation procedure

LIMITATIONS AND CAVEATS:
Study terminated early due to clinical equipoise

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT02324465/Prot_SAP_000.pdf